CLINICAL TRIAL: NCT06781710
Title: Retrospective Analysis of the Epidemiology, Clinical Presentation and Therapy as Well as Therapy-associated Risk of Demyelination Syndrome in Patients With Profound Hyponatremia in the Emergency Department
Brief Title: Analysis of the Epidemiology, Clinical Presentation and Therapy as Well as Therapy-associated Risk of Demyelination Syndrome in Patients With Profound Hyponatremia in the Emergency Department
Acronym: ProfHN_in_ZNA
Status: Recruiting | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Volker Burst, Prof. Dr. med., University of Cologne
Other Study IDs: V1.0_23.09.2022; 22-1373-retro (Other: Ethics Committee)
Record Dates: First submitted 2024-12-17; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Hyponatremia
Keywords: Hyponatremia; ODS; demyelination; overcorrection
MeSH Terms: conditions — Hyponatremia; Demyelinating Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hyponatremia is a frequent cause for presentation to the emergency department (ED). While patients with chronic hyponatremia often exhibit minor symptoms, acute development of hyponatremia can lead to global cerebral edema, transtentorial herniation and death. The time course of hyponatremia development is usually not known to the treating physician at presentation. Hence, type and extent of therapy depend on the presence or absence of severe symptoms such as coma, seizures, obtundation or vomiting. It is believed that these are suggestive of increased cerebral pressure and indicative of cerebral edema. International guidance thus demands aggressive therapy with hypertonic saline at their occurrence. However, severe symptoms can also be found in patients with chronic hyponatremia (i.e., development in more than 48 hours) which are not at risk for developing cerebral edema due to adaptive counter measures in the brain. Although the percentage of patients with severe symptoms in chronic hyponatremia is considerably smaller than in acute hyponatremia, a higher incidence of chronic hyponatremia may lead to a larger overall number of severely symptomatic patients with chronic hyponatremia. The precise distribution of acute and chronic cases in the ED has not been established yet. In consequence, many patients with hyponatremia presenting with severe symptoms receive aggressive treatment in order to raise sodium levels, exposing them to the risk for overly rapid correction and osmotic demyelination syndrome (ODS). Current U.S. recommendations limit the sodium increase to a maximum of 8 mmol/L and 10-12 mmol/L in the first 24 hours in patients with high or low-to-moderate ODS risk, respectively. Similarly, the 2014 European Clinical Practice Guideline (ECPG) recommends a limit of 10 mmol/L in each 24h-period. These limits are often not accomplished in the real-world setting. In summary, weighing the risk of hyponatremia against complications associated with its (over-)correction constitutes a dilemma for the clinician. It will be strived to refine guidance on management of hyponatremia in patients with profound hyponatremia. Therefore, a better understanding of the proportions and characteristics of patients at risk for both cerebral edema and ODS is needed. The primary objective of this study is to determine the rate of hyponatremic patients who had already developed cerebral edema on admission and to identify patients who developed ODS during the index hospital stay. A secondary objective is a more detailed characterization of these subsets.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years
* Plasma sodium ≤125 mmol/L in the initial blood sample after admission to the Emergency Department

Exclusion Criteria:

* Lack of follow-up sodium analyses within the first 24 hours after admission
* initial blood glucose >300 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with profound hyponatremia presenting to the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with cerebral edema | on admission and within 2 hours after admission
  The primary aim is to determine the patient´s risk to develop cerebral edema, associated with hyponatremia and osmotic demyelination as a result of therapy, respectively.
  Determination at admission as evidenced by imaging studies in the time period index admission in the Emergency Department until referral from the Emergency Department
rate of patients who develop osmotic demyelination syndrome (ODS) | on admission and 90 days after admission
  The primary aim is to determine the patient´s risk to develop cerebral edema, associated with hyponatremia and osmotic demyelination as a result of therapy, respectively.
  Determination as evidenced by imaging studies in the time period index admission until 90 days thereafter.

SECONDARY OUTCOMES:
Risk factors associated with hyponatremia | on admission
  Are there specific risk factors apart from hyponatremia or its management that influence the development of cerebral edema, respectively?
Risk factors associated with osmotic demyelination syndrome | on admission
  Are there specific risk factors apart from hyponatremia or its management that influence the development of osmotic demyelination syndrome, respectively?
Proportion of patients with severe symptoms and characterization of severe symptoms of hyponatremia | on admission
  Determine the rate of patients with profound hyponatremia that exhibit severe symptoms such as vomiting, obtundation, seizures, coma and cardiorespiratory distress.
Proportion of patients, in which ODS was considered "confirmed", "highly likely" and "possible", considering clinical and/or radiological features of ODS | at study end, 1 year after study start
  Determine the rate of patients, in which ODS was considered "confirmed" in patients with classical radiological findings, "highly likely" in patients with clinical features of and radiological findings consistent with ODS, and "possible" in patients with clinical but no radiological features (or that had not received imaging)

CONTACTS AND LOCATIONS:
Overall Officials: Volker Burst, MD, Principal Investigator — University Hospital Cologne
Locations (1):
- University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No
Data base will be shared upon request